CLINICAL TRIAL: NCT02176837
Title: Evaluation of Intravenous Nitrite Infusion for Reversal of Cerebral Vasospasm After Subarachnoid Hemorrhage From a Cerebral Aneurysm
Brief Title: Intravenous Nitrite Infusion for Reversal of Cerebral Vasospasm After Subarachnoid Hemorrhage
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Hope Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SN-03-01
Record Dates: First submitted 2014-02-19; First posted 2014-06-27 (Estimated); Results first posted 2018-02-08 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Subarachnoid Hemorrhage
Keywords: subarachnoid hemorrhage; vasospasm; nitrite; sodium nitrite
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Sodium Nitrite

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sodium Nitrite (Experimental): One dose cohort is planned, 64 nmol/min/kg sodium nitrite (0.1325 mg/hour/kg; 0.0442 ml/hour/kg at a concentration of 3mg/ml).
  Interventions: Drug: Sodium Nitrite

INTERVENTIONS:
Drug: Sodium Nitrite — Subjects will receive continuous intravenous infusion of study drug for 7 days at a dose of 64 nmol/min/kg. The infusion will begin shortly after angiographic demonstration of cerebral vasospasm and will be for 7 days unless side effects of the drug dictate stopping the infusion.
  Other Names: Sodium Nitrite Injection 300 mg/10 mL

SUMMARY:
The hypothesis is that intravenous infusion of sodium nitrite is safe and effective for the reversal of cerebral vasospasm after subarachnoid hemorrhage in patients with a cerebral aneurysm.

DETAILED DESCRIPTION:
This is a pilot single center, open-labeled study. Patients with subarachnoid hemorrhage admitted to the hospital and who meet entry criteria will be offered enrollment into the study. The patients will be enrolled promptly after detection of the presence of cerebral vasospasm. Subjects will receive sodium nitrite infusion.

One dose cohort is planned, 64 nmol/min/kg sodium nitrite (0.1325 mg/hour/kg; 0.0442 ml/hour/kg at a concentration of 3mg/ml).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained from a patient or legal representative before enrollment;
* Admission to hospital following subarachnoid hemorrhage;
* Aneurysm confirmed by digital subtraction angiography or CT-angiography after admission;
* Development of the clinical symptoms and /or signs of cerebral vasospasm and CT-angiography results warranting cerebral angiography.

Exclusion Criteria:

* Rupture of a fusiform, traumatic, or mycotic aneurysm;
* Pregnancy (confirmed by a serum human chorionic gonadotropin pregnancy test) or breast feeding;
* Methemoglobin > 2%
* History of sickle cell disease, thalassemia, or other hemoglobinopathy;
* Anemia with hemoglobin level less than 6 g/dL;
* Significant acute or chronic concomitant diseases (including renal, hepatic, cardiovascular, pulmonary, or oncologic disease, sepsis, pulmonary edema, pulmonary embolism) that would be inconsistent with survival for at least 6 months;
* History of allergy to nitrites or allergy to other substances that could interfere with nitrite metabolism, within 30 days before screening;
* History of red blood cell glucose-6-phosphate dehydrogenase (G6PD)deficiency;
* Treatment with allopurinol, a medication that could interfere with nitrite metabolism, within 30 days before screening;
* Other investigational drug within the past 30 days;
* other cerebral injury within the past 30 days including previous subarachnoid hemorrhage, stroke, transient ischemic attacks (TIA), concussion, head trauma, cranial surgery, radiation therapy to the head.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-06; Primary Completion 2017-01-15 (Actual); Study Completion 2017-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenny Liu, MD, Principal Investigator — University of Virginia Medical Center, Department of Neurosurgery
Locations (1):
- University of Virginia Medical Center, Charlottesville, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sodium Nitrite: 64 nmol/min/kg sodium nitrite
Period: Overall Study
Arm/Group | Sodium Nitrite
Started | 6
Completed | 0
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Sodium Nitrite
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Cerebral Vasospasm
Description: Cerebral digital subtraction angiographies will be reviewed at at least 2 time points, including at the time of diagnosis of angiographic vasospasm immediately before treatment with nitrite and after up to 180 minutes of nitrite infusion. Radiographs will be compared to determine whether increased flow of radiographic dye is visualized following initiation of nitrite infusion.
Time Frame: 180 minutes
Population: Patients who received sodium nitrite
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Nitrite
Number analyzed (Participants) | 6
Participants
  Increased flow between baseline and 2nd radiograph | 2
  Unchanged flow between baseline and 2nd radiograph | 4

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Regular investigator assessment
Arm/Group | Sodium Nitrite
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No